CLINICAL TRIAL: NCT02927769
Title: Risk-based, Response-adapted, Phase II Open-label Trial of Nivolumab + Brentuximab Vedotin (N + Bv) for Children, Adolescents, and Young Adults With Relapsed/Refractory (R/R) CD30 + Classic Hodgkin Lymphoma (cHL) After Failure of First-line Therapy, Followed by Brentuximab + Bendamustine (Bv + B) for Participants With a Suboptimal Response (CheckMate 744: CHECKpoint Pathway and Nivolumab Clinical Trial Evaluation)
Brief Title: A Study of Nivolumab Plus Brentuximab Vedotin in Patients Between 5 and 30 Years Old, With Hodgkin's Lymphoma (cHL), Relapsed or Refractory From First Line Treatment
Acronym: CheckMate 744
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-744; 2016-002347-41 (EudraCT Number)
Expanded Access: NCT02475382 (No longer available)
Record Dates: First submitted 2016-10-06; First posted 2016-10-07 (Estimated); Results first posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Hodgkin Disease
MeSH Terms: conditions — Hodgkin Disease | interventions — Nivolumab; Brentuximab Vedotin; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nivolumab + brentuximab vedotin (Experimental)
  Interventions: Biological: Nivolumab; Biological: brentuximab vedotin
- brentuximab vedotin + bendamustine (Experimental)
  Interventions: Biological: brentuximab vedotin; Biological: bendamustine

INTERVENTIONS:
Biological: Nivolumab — Specified Dose on Specified Days
  Other Names: BMS-936558; Opdivo
  Arms: Nivolumab + brentuximab vedotin
Biological: brentuximab vedotin — Specified Dose on Specified Days
Biological: bendamustine — Specified Dose on Specified Days
  Arms: brentuximab vedotin + bendamustine

SUMMARY:
The purpose of this study is to determine whether nivolumab plus brentuximab vedotin (followed by brentuximab vedotin plus bendamustine in patient with suboptimal response) is safe and effective in treating patients with Hodgkin's lymphoma (cHL). Eligible patients are children, adolescents, and young adults relapsed or refractory to first line.

ELIGIBILITY:
Inclusion Criteria:

* Classic Hodgkin Lymphoma (cHL), relapsed or refractory
* Minimal limitation on activities of daily living as measured by Karnofsky ≥ 50 for participants > 16 years of age or Lansky ≥ 50 for participants ≤ 16 years of age.
* One prior anti-cancer therapy that did not work

Exclusion Criteria:

* Active, known, or suspected autoimmune disease or infection
* Active cerebral/meningeal disease related to the underlying malignancy
* More than one line of anti-cancer therapy or no treatment at all
* Received a stem cell transplant for Hodgkin Lymphoma and/or a solid organ transplant
* Prior treatment with any drug that targets T cell co-stimulation pathways (such as checkpoint inhibitors)

Other protocol defined inclusion/exclusion criteria apply

Ages: 5 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 72 (Actual)
Dates: Start 2017-03-28 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (79):
- United States (43):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Phoenix Children'S Hospital, Phoenix, Arizona
  - Loma Linda University Cancer Center, Loma Linda, California
  - Valley Children's Hospital, Madera, California
  - Children'S Hospital & Research Center At Oakland, Oakland, California
  - Children'S Hospital Of Orange County, Orange, California
  - Lucile Packard Children'S Research Hospital/Stanford Univ, Palo Alto, California
  - Local Institution - 0091, San Diego, California
  - Childrens Hospital of Colorado, Aurora, Colorado
  - Smilow Cancer Hospital At Yale New Haven Hospital, New Haven, Connecticut
  - Nemours / A. I. duPont Hospital for Children, Wilmington, Delaware
  - Children'S National Medical Center, Washington D.C., District of Columbia
  - Local Institution - 0062, Jacksonville, Florida
  - Local Institution - 0069, St. Petersburg, Florida
  - Children's Healthcare Of Atlanta, Atlanta, Georgia
  - University Of Iowa, Iowa City, Iowa
  - Local Institution - 0070, Baltimore, Maryland
  - Dana Farber Cancer Institute., Boston, Massachusetts
  - Local Institution - 0097, Detroit, Michigan
  - Local Institution - 0049, Jackson, Mississippi
  - Local Institution - 0085, Kansas City, Missouri
  - Washington University School Of Medicine, St Louis, Missouri
  - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Local Institution - 0067, Hackensack, New Jersey
  - Local Institution - 0047, New Brunswick, New Jersey
  - Local Institution - 0068, Buffalo, New York
  - Local Institution, Chapel Hill, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Cincinnati Children'S Hospital Medical Center, Cincinnati, Ohio
  - Local Institution - 0089, Columbus, Ohio
  - University Of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Local Institution - 0090, Hershey, Pennsylvania
  - Childrens Hospital Of Philadelphia, Philadelphia, Pennsylvania
  - Childrens Hospital Of Pittsburgh Of Upmc, Pittsburgh, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - Local Institution - 0042, Austin, Texas
  - Local Institution - 0071, Dallas, Texas
  - Baylor College Of Medicine, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Children'S Hosp-Kings Daughter, Norfolk, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Local Institution - 0048, Seattle, Washington
  - Local Institution - 0065, Milwaukee, Wisconsin
- Canada (3):
  - Local Institution, Calgary, Alberta
  - Local Institution - 0092, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
- Klinika detske hematologie a onkologie, Prague, Czechia
- France (9):
  - Local Institution - 0034, Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - Local Institution - 0030, Lille
  - Local Institution - 0029, Lyon
  - Local Institution - 0032, Marseille
  - Local Institution - 0028, Nantes
  - Local Institution - 0031, Paris
  - Local Institution - 0026, Paris
  - Local Institution - 0033, Toulouse
  - Local Institution - 0027, Villejuif
- Germany (4):
  - Local Institution - 0056, Berlin
  - Local Institution - 0055, Giessen
  - Local Institution - 0057, Hanover
  - Local Institution - 0102, München
- Local Institution - 0017, Dublin, Ireland
- Italy (6):
  - Local Institution - 0024, Aviano (PN)
  - Local Institution - 0020, Bologna
  - Local Institution - 0021, Genova
  - Local Institution - 0019, Monza (mb)
  - Local Institution - 0023, Napoli
  - Local Institution - 0022, Roma
- Netherlands (2):
  - Local Institution - 0001, Rotterdam
  - Local Institution - 0006, Utrecht
- Poland (2):
  - Local Institution, Gdansk
  - Local Institution, Krakow
- Spain (2):
  - Local Institution - 0082, Barcelona
  - Local Institution - 0084, Madrid
- United Kingdom (6):
  - Local Institution - 0035, Leeds, North Yorkshire
  - Local Institution, Leeds, Yorkshire
  - Local Institution, Birmingham
  - Local Institution, Glasgow
  - Local Institution - 0002, London
  - Local Institution - 0012, Manchester

REFERENCES:
- [Derived] Daw S, Cole PD, Hoppe BS, Hodgson D, Beishuizen A, Garnier N, Buffardi S, Mascarin M, Lissat A, Mauz-Korholz C, Krajewski J, Akyol A, Crowe R, Anderson B, Xu Y, Drachtman RA, Kelly KM, Leblanc T, Harker-Murray P. Transplant-Free Approach in Relapsed Hodgkin Lymphoma in Children, Adolescents, and Young Adults: A Nonrandomized Clinical Trial. JAMA Oncol. 2025 Mar 1;11(3):249-257. doi: 10.1001/jamaoncol.2024.5627. PMID 39745739
- [Derived] Harker-Murray P, Mauz-Korholz C, Leblanc T, Mascarin M, Michel G, Cooper S, Beishuizen A, Leger KJ, Amoroso L, Buffardi S, Rigaud C, Hoppe BS, Lisano J, Francis S, Sacchi M, Cole PD, Drachtman RA, Kelly KM, Daw S. Nivolumab and brentuximab vedotin with or without bendamustine for R/R Hodgkin lymphoma in children, adolescents, and young adults. Blood. 2023 Apr 27;141(17):2075-2084. doi: 10.1182/blood.2022017118. PMID 36564047
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants entered the Induction phase and received treatment with nivolumab + brentuximab vedotin (N+ Bv) Participants moved into the Intensification phase if they received treatment with brentuximab + bendamustine (Bv + B).
  Participants moved into the Consolidation Phase if they received radiation therapy (Cohort 1) or high-dose chemotherapy followed by an autologous stem cell transplant (HDCT/ASCT) (Cohort 2).
Groups:
- Cohort 1: Relapsed/Refractory Classic Hodgkin Lymphoma - Low Risk Relapse: Participants started in the induction phase and received nivolumab + brentuximab vedotin (N+Bv) for 2 cycles (6 weeks). Participants with radiographic progression, as assessed by Investigator at Cycle 2 entered follow-up. The rest of the participants continued in the induction phase and received 2 additional cycles of N+Bv study therapy (total 4 cycles = 12 weeks).
  * Participants who had a complete metabolic response (CMR) by BICR after a total of 4 cycles (12 weeks) of N+Bv received an additional 2 cycles of treatment of N+Bv (for a total of 6 cycles [18 weeks]), followed by Radiation Therapy (RT) (consolidation phase).
  * Participants without a CMR after 4 cycles of N+Bv, by BICR, entered the intensification phase and received 2 cycles of brentuximab + bendamustine (Bv+B); participants who achieved CMR after these 2 cycles proceeded with RT (consolidation phase).
  * Participants who had radiographic progression after Cycle 4 N+Bv, as assessed by BICR, or those who did not achieve CMR, by BICR, after 2 cycles of Bv+B were taken off study treatment and entered follow-up.
- Cohort 2: Relapsed/Refractory Classic Hodgkin Lymphoma - Standard Risk Relapse: Participants started in the induction phase and received nivolumab + brentuximab vedotin (N+Bv) for 2 cycles (6 weeks). Participants with radiographic progression, as assessed by Investigator at Cycle 2 entered follow-up. The rest of the participants received 2 additional cycles of N+Bv study therapy (total 4 cycles = 12 weeks).
  * Participants who had complete metabolic response (CMR), by BICR, after a total of 4 cycles (12 weeks) of N+Bv proceeded with high-dose chemotherapy followed by an autologous stem cell transplant (HDCT/ASCT) (consolidation phase). Participants with CMR had the option to receive up to 2 additional cycles of N+Bv if their HDCT/ASCT was postponed for any reason.
  * Participants without a CMR, by BICR, after 4 cycles of N+Bv received 2 cycles of brentuximab + bendamustine (Bv+B) (intensification phase).
  * Participants in CMR, by BICR, after 2 cycles of Bv+B received HDCT/ASCT (consolidation phase).
  * Participants without CMR by BICR could receive 2 additional cycles of Bv+B. If these participants attained CMR, they proceeded with HDCT/ASCT (consolidation phase).
  * Participants with CMR had the option to receive up to 2 additional cycles of B+Bv if their HDCT/ASCT was postponed.
  * Participants who had radiographic progression after Cycle 4 N+Bv, during study treatment or those who did not achieve CMR after final cycle of Bv+B were taken off study treatment and entered follow-up.
Period: Induction Phase
Arm/Group | Cohort 1: Relapsed/Refractory Classic Hodgkin Lymphoma - Low Risk Relapse | Cohort 2: Relapsed/Refractory Classic Hodgkin Lymphoma - Standard Risk Relapse
Started | 28 | 44
Completed | 27 | 42
Not Completed | 1 | 2
Not completed — Study drug toxicity | 1 | 1
Not completed — Disease progression | 0 | 1
Period: Consolidation Phase
Arm/Group | Cohort 1: Relapsed/Refractory Classic Hodgkin Lymphoma - Low Risk Relapse | Cohort 2: Relapsed/Refractory Classic Hodgkin Lymphoma - Standard Risk Relapse
Started | 22 | 32
Completed | 22 | 32
Not Completed | 0 | 0
Period: Intensification Phase
Arm/Group | Cohort 1: Relapsed/Refractory Classic Hodgkin Lymphoma - Low Risk Relapse | Cohort 2: Relapsed/Refractory Classic Hodgkin Lymphoma - Standard Risk Relapse
Started | 6 | 11
Completed | 5 | 11
Not Completed | 1 | 0
Not completed — Study drug toxicity | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Relapsed/Refractory Classic Hodgkin Lymphoma - Low Risk Relapse | Cohort 2: Relapsed/Refractory Classic Hodgkin Lymphoma - Standard Risk Relapse | Total
Number analyzed (Participants) | 28 | 44 | 72
Age, Continuous [Mean (Standard Deviation); unit: Years] | 17.0 (4.3) | 16.2 (3.7) | 16.5 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 15 | 33
  Male | 10 | 29 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 8 | 20 | 28
  Unknown or Not Reported | 17 | 23 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 1 | 1 | 2
  White | 25 | 41 | 66
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Complete Metabolic Response (CMR) Rate at Any Time Prior to Radiation Therapy by Blinded Independent Centralized Review (BICR) - Cohort 1
Description: The complete metabolic response (CMR) rate is defined as the percent of all response-evaluable participants who, assessed by the BICR, achieved best response of CMR.
  Complete metabolic response (CMR):
  * Lymph nodes/extralymphatic sites: Score 1, 2, 3 with/without residual mass on 5-point scale
  * New lesions: No
  * Bone marrow: No FDG-avid disease Participants who stopped study treatment early for toxicity without a CMR were evaluable.
  Confidence interval is based on the Clopper and Pearson method
Time Frame: From first dose to complete metabolic response or the completion of six cycles of therapy (up to approximately 18 weeks).
Population: All treated participants in Cohort 1. Prespecified to be collected for Cohort 1 only.
Measure: Number (90% Confidence Interval); unit: Percent of participants
Arm/Group | Cohort 1: Relapsed/Refractory Classic Hodgkin Lymphoma - Low Risk Relapse
Number analyzed (Participants) | 28
Percent of participants | 92.9 [79.2 to 98.7]

2. Primary Outcome: Event-free Survival (EFS) Rate at 3 Years by Blinded Independent Centralized Review (BICR) - Cohort 1
Description: Event Free Survival (EFS) is the time from the first treatment to the earliest occurrence of composite events including: Disease progression (PD), Failure to achieve complete metabolic response (CMR) after 4 cycles of N+Bv and 2 cycles of Bv+B, Secondary malignancy, Death .
  PD :
  Lymph Nodes and Lesions: new growth or increase of >= 50% in size from nadir. New or growing lesions outside the lymph nodes.
  Spleen: Significant increase in spleen size, either from a previously enlarged state or from normal size.
  New Lesions: Yes Bone Marrow: New or returning FDG-avid disease
  CMR:
  Lymph nodes/extralymphatic sites: Score 1, 2, 3 with/without residual mass on 5-point scale New lesions: No Bone marrow: No FDG-avid disease Participants without an "event" were censored at the last tumor assessment. Those who started subsequent anticancer therapy without a prior "event" were censored at the last tumor assessment prior to or upon starting subsequent therapy.
  Based on Kaplan-Meier Estimates.
Time Frame: At 3 years post first dose of study therapy
Population: All treated participants in Cohort 1. Prespecified to be collected for Cohort 1 only.
Measure: Number (90% Confidence Interval); unit: Percent of participants
Arm/Group | Cohort 1: Relapsed/Refractory Classic Hodgkin Lymphoma - Low Risk Relapse
Number analyzed (Participants) | 28
Percent of participants | 87.5 [70.6 to 95.0]

3. Primary Outcome: Complete Metabolic Response (CMR) Rate at Any Time Prior to High Dose Chemotherapy Followed by Autologous Stem Cell Treatment (HDCT/ASCT) by Blinded Independent Centralized Review (BICR) - Cohort 2
Description: The complete metabolic response (CMR) rate is defined as the percent of all response-evaluable participants who, assessed by the BICR, achieved best response of CMR.
  Complete metabolic response (CMR):
  * Lymph nodes/extralymphatic sites: Score 1, 2, 3 with/without residual mass on 5-point scale
  * New lesions: No
  * Bone marrow: No FDG-avid disease Participants who came off study treatment early for toxicity without a CMR were evaluable.
  Confidence interval is based on the Clopper and Pearson method
Time Frame: as for outcome 1
Population: All treated participants in Cohort 2. Prespecified to be collected for Cohort 2 only.
Measure: Number (90% Confidence Interval); unit: Percent of participants
Arm/Group | Cohort 2: Relapsed/Refractory Classic Hodgkin Lymphoma - Standard Risk Relapse
Number analyzed (Participants) | 44
Percent of participants | 88.6 [77.6 to 95.4]

4. Secondary Outcome: Overall Response Rate (ORR) Following 4 Cycles of Nivolumab + Brentuximab Vedotin Treatment by Blinded Independent Centralized Review (BICR)
Description: Overall response rate (ORR) is defined as the percent of all response-evaluable participants who, assessed by the BICR, achieved a best response of complete metabolic response (CMR) or partial metabolic response (PMR).
  Complete metabolic response (CMR):
  * Lymph nodes/extralymphatic sites: Score 1, 2, 3 with/without residual mass on 5-point scale
  * New lesions: No
  * Bone marrow: No FDG-avid disease
  Partial metabolic response (PMR):
  * Lymph nodes/extralymphatic: Score 4 or 5, reduced uptake from baseline
  * New lesions: None
  * Bone marrow: Residual uptake higher than normal, reduced from baseline. Participants who came off early for toxicity without CMR or PMR were evaluable.
Time Frame: From first dose to PMR or CMR within 4 cycles of therapy, or the completion of four cycles of therapy (N+Bv x4) (up to approximately 12 weeks).
Population: All treated participants.
Measure: Number (90% Confidence Interval); unit: Percent of participants
Arm/Group | Cohort 1: Relapsed/Refractory Classic Hodgkin Lymphoma - Low Risk Relapse | Cohort 2: Relapsed/Refractory Classic Hodgkin Lymphoma - Standard Risk Relapse
Number analyzed (Participants) | 28 | 44
Percent of participants | 96.4 [84.1 to 99.8] | 93.2 [83.3 to 98.1]

5. Secondary Outcome: Progression Free Survival (PFS) Rate at 3 Years by Blinded Independent Centralized Review (BICR)
Description: Progression Free Survival (PFS) is the time from the date of first treatment to the date of first documented disease progression by BICR or death.
  Progressive Disease (PD):
  Lymph Nodes and Lesions: new growth or increase of >= 50% in size from nadir. New or growing lesions outside the lymph nodes.
  Spleen: Significant increase in spleen size, either from a previously enlarged state or from normal size.
  New Lesions: Yes Bone Marrow: New or returning FDG-avid disease. Participants who neither progressed nor died were censored at the last adequate tumor assessment. Participants who started subsequent anticancer therapy (that is not part of high dose chemotherapy followed by autologous stem cell transplant (HDCT/ASCT) Consolidation Therapy for R2 Cohort) without a prior reported progression or death were censored at the last tumor assessment prior to initiation of the subsequent anticancer therapy.
  Based on Kaplan-Meier Estimates.
Time Frame: At 3 years post first dose of study therapy
Population: All treated participants.
Measure: Number (90% Confidence Interval); unit: Percent of participants
Arm/Group | Cohort 1: Relapsed/Refractory Classic Hodgkin Lymphoma - Low Risk Relapse | Cohort 2: Relapsed/Refractory Classic Hodgkin Lymphoma - Standard Risk Relapse
Number analyzed (Participants) | 28 | 44
Percent of participants | 95.2 [77.7 to 99.1] | 91.1 [78.4 to 96.5]

6. Secondary Outcome: Duration of Response (DOR) by Blinded Independent Centralized Review (BICR)
Description: Duration of response (DOR) is the time from first complete metabolic response or partial metabolic response (CMR or PMR) to event free survival EFS (Cohort 1)/progression free survival PFS (Cohort 2) event. For participants with no event, DOR was censored on the date of last tumor assessment.
  Participants who started subsequent anticancer therapy (not part of high-dose chemotherapy followed by autologous stem cell transplant HDCT/ASCT) without a prior reported EFS/PFS event were censored at the last tumor assessment prior to initiation of the subsequent therapy.
  Complete metabolic response (CMR):
  * Lymph nodes/extralymphatic sites: Score 1, 2, 3 with/without residual mass on 5-point scale
  * New lesions: No
  * Bone marrow: No FDG-avid disease
  Partial metabolic response (PMR):
  * Lymph nodes/extralymphatic: Score 4 or 5, reduced uptake from baseline
  * New lesions: None
  * Bone marrow: Residual uptake higher than normal, reduced from baseline. Based on Kaplan-Meier estimates
Time Frame: From first dose until disease progression, start of subsequent anti-cancer therapy, or or death due to any cause (up to approximately 86 months)
Population: All treated participants with a response of complete metabolic response (CMR) or partial metabolic response (PMR).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1: Relapsed/Refractory Classic Hodgkin Lymphoma - Low Risk Relapse | Cohort 2: Relapsed/Refractory Classic Hodgkin Lymphoma - Standard Risk Relapse
Number analyzed (Participants) | 28 | 43
Months | NA [NA to NA] — Insufficient number of events to calculate median or confidence interval using Kaplan-Meier estimates. | NA [NA to NA] — Insufficient number of events to calculate median or confidence interval using Kaplan-Meier estimates.

7. Secondary Outcome: Complete Metabolic Response (CMR) Rate at Any Time Prior to Radiation Therapy by Investigator - Cohort 1
Description: The complete metabolic response (CMR) rate is defined as the percent of all response-evaluable participants who, assessed by the investigator, achieved best response of CMR.
  Complete metabolic response (CMR):
  * Lymph nodes/extralymphatic sites: Score 1, 2, 3 with/without residual mass on 5-point scale
  * New lesions: No
  * Bone marrow: No FDG-avid disease Participants who come off early for toxicity without a CMR were evaluable. Confidence interval is based on the Clopper and Pearson method
Time Frame: as for outcome 1
Population: All treated participants in Cohort 1. Prespecified to be collected for Cohort 1 only.
Measure: Number (90% Confidence Interval); unit: Percent of participants
Arm/Group | Cohort 1: Relapsed/Refractory Classic Hodgkin Lymphoma - Low Risk Relapse
Number analyzed (Participants) | 28
Percent of participants | 89.3 [74.6 to 97.0]

8. Secondary Outcome: Event-free Survival (EFS) Rate at 3 Years by Investigator - Cohort 1
Description: as for outcome 2
Time Frame: At 3 years post first dose of study therapy
Population: All treated participants in Cohort 1. Prespecified to be collected for Cohort 1 only.
Measure: Number (90% Confidence Interval); unit: Percent of participants
Arm/Group | Cohort 1: Relapsed/Refractory Classic Hodgkin Lymphoma - Low Risk Relapse
Number analyzed (Participants) | 28
Percent of participants | 88.5 [72.8 to 95.4]

9. Secondary Outcome: Complete Metabolic Response (CMR) Rate at Any Time Prior to High Dose Chemotherapy Followed by Autologous Stem Cell Treatment (HDCT/ASCT) by Investigator - Cohort 2
Description: The complete metabolic response (CMR) rate is defined as the percent of all response-evaluable participants who, assessed by the investigator, achieved best response of CMR.
  Complete metabolic response (CMR):
  * Lymph nodes/extralymphatic sites: Score 1, 2, 3 with/without residual mass on 5-point scale
  * New lesions: No
  * Bone marrow: No FDG-avid disease Participants who came off study treatment early for toxicity without a CMR were evaluable.
  Confidence interval is based on the Clopper and Pearson method.
Time Frame: as for outcome 1
Population: All treated participants in Cohort 2. Prespecified to be collected for Cohort 2 only.
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Cohort 2: Relapsed/Refractory Classic Hodgkin Lymphoma - Standard Risk Relapse
Number analyzed (Participants) | 44
Percent of participants | 86.4 [74.8 to 93.9]

10. Secondary Outcome: Overall Response Rate (ORR) Following 4 Cycles of Nivolumab + Brentuximab Vedotin Treatment by Investigator
Description: Overall response rate (ORR) is defined as the percent of all response-evaluable participants who, assessed by the investigator, achieve a best response of complete metabolic response (CMR) or partial metabolic response (PMR).
  Complete metabolic response (CMR):
  * Lymph nodes/extralymphatic sites: Score 1, 2, 3 with/without residual mass on 5-point scale
  * New lesions: No
  * Bone marrow: No FDG-avid disease
  Partial metabolic response:
  * Lymph nodes/extralymphatic: Score 4 or 5, reduced uptake from baseline
  * New lesions: None
  * Bone marrow: Residual uptake higher than normal, reduced from baseline Participants who came off early for toxicity without CMR or PMR were evaluable.
Time Frame: as for outcome 4
Population: All treated participants.
Measure: Number (90% Confidence Interval); unit: Percent of participants
Arm/Group | Cohort 1: Relapsed/Refractory Classic Hodgkin Lymphoma - Low Risk Relapse | Cohort 2: Relapsed/Refractory Classic Hodgkin Lymphoma - Standard Risk Relapse
Number analyzed (Participants) | 28 | 44
Percent of participants | 100.0 [89.9 to 100.0] | 90.9 [80.4 to 96.8]

11. Secondary Outcome: Progression Free Survival (PFS) Rate at 3 Years by Investigator
Description: Progression Free Survival (PFS) is the time from the date of first treatment to the date of first documented disease progression by investigator or death.
  Progressive Disease (PD):
  Lymph Nodes and Lesions: new growth or increase of >= 50% in size from nadir. New or growing lesions outside the lymph nodes.
  Spleen: Significant increase in spleen size, either from a previously enlarged state or from normal size.
  New Lesions: Yes Bone Marrow: New or returning FDG-avid disease. Participants who neither progressed nor died were be censored at the last adequate tumor assessment. Participants who started subsequent anticancer therapy (that is not part of high dose chemotherapy followed by autologous stem cell transplant (HDCT/ASCT) Consolidation Therapy forR2 Cohort) without a prior reported progression or death were censored at the last tumor assessment prior to initiation of the subsequent anticancer therapy.
  Based on Kaplan-Meier Estimates.
Time Frame: At 3 years post first dose
Population: All treated participants.
Measure: Number (90% Confidence Interval); unit: Percent of participants
Arm/Group | Cohort 1: Relapsed/Refractory Classic Hodgkin Lymphoma - Low Risk Relapse | Cohort 2: Relapsed/Refractory Classic Hodgkin Lymphoma - Standard Risk Relapse
Number analyzed (Participants) | 28 | 44
Percent of participants | 95.8 [80.2 to 99.2] | 88.1 [74.8 to 94.6]

12. Secondary Outcome: Duration of Response (DOR) by Investigator
Description: Duration of response (DOR) is the time from first complete metabolic response or partial metabolic response (CMR or PMR) to event free survival EFS (Cohort 1)/progression free survival PFS (Cohort 2) event. For participants with no event, the DOR was censored on the date of last tumor assessment.
  Participants who started subsequent anticancer therapy (not part of high-dose chemotherapy followed by autologous stem cell transplant HDCT/ASCT) without a prior reported EFS/PFS event were censored at the last tumor assessment prior to initiation of the subsequent anticancer therapy.
  Complete metabolic response (CMR):
  * Lymph nodes/extralymphatic sites: Score 1, 2, 3 with/without residual mass on 5-point scale
  * New lesions: No
  * Bone marrow: No FDG-avid disease
  Partial metabolic response:
  * Lymph nodes/extralymphatic: Score 4 or 5, reduced uptake from baseline
  * New lesions: None
  * Bone marrow: Residual uptake higher than normal, reduced from baseline. Based on Kaplan-Meier estimates.
Time Frame: as for outcome 6
Population: All treated participants with a response of complete metabolic response (CMR) or partial metabolic response (PMR).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1: Relapsed/Refractory Classic Hodgkin Lymphoma - Low Risk Relapse | Cohort 2: Relapsed/Refractory Classic Hodgkin Lymphoma - Standard Risk Relapse
Number analyzed (Participants) | 28 | 44
Months | NA [NA to NA] — Insufficient number of events to calculate median or confidence interval using Kaplan-Meier estimates. | NA [NA to NA] — Insufficient number of events to calculate median or confidence interval using Kaplan-Meier estimates.

13. Secondary Outcome: The Number of Participants With Adverse Events (AEs)
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study drug and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (such as an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug.
Time Frame: From first dose to 30 days post last dose (an average of 4 months up until a maximum of 7 months).
Population: All treated participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Relapsed/Refractory Classic Hodgkin Lymphoma - Low Risk Relapse | Cohort 2: Relapsed/Refractory Classic Hodgkin Lymphoma - Standard Risk Relapse
Number analyzed (Participants) | 28 | 44
Participants | 26 | 42

14. Secondary Outcome: The Number of Participants With Serious Adverse Events (SAEs)
Description: A Serious Adverse Event (SAE) is defined as any untoward medical occurrence that, at any dose:
  * Results in death
  * Is life-threatening (defined as an event in which the participant was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe)
  * Requires inpatient hospitalization or causes prolongation of existing hospitalization
  * Results in persistent or significant disability/incapacity
  * Is a congenital anomaly/birth defect
  * Is an important medical event.
Time Frame: From first dose to 30 days post last dose (an average of 4 months up until a maximum of 7 months)
Population: All treated participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Relapsed/Refractory Classic Hodgkin Lymphoma - Low Risk Relapse | Cohort 2: Relapsed/Refractory Classic Hodgkin Lymphoma - Standard Risk Relapse
Number analyzed (Participants) | 28 | 44
Participants | 8 | 9

15. Secondary Outcome: The Number of Participants With Abnormal Laboratory Values for Specific Thyroid Tests
Description: The Number of Participants with Abnormal Laboratory Values for Specific Thyroid Tests.
Time Frame: From first dose to 30 days post last dose (an average of 4 months up until a maximum of 7 months)
Population: All treated participants with at least one on treatment TSH measurement.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Relapsed/Refractory Classic Hodgkin Lymphoma - Low Risk Relapse | Cohort 2: Relapsed/Refractory Classic Hodgkin Lymphoma - Standard Risk Relapse
Number analyzed (Participants) | 28 | 44
Participants
  TSH > ULN | 6 | 8
  TSH > ULN WITH TSH <= ULN AT BASELINE | 5 | 4
  TSH >ULN WITH ATLEAST ONE FT3/FT4 TEST VALUE <LLN | 1 | 0
  TSH >ULN WITH ALL OTHER FT3/FT4 TEST VALUES >= LLN | 4 | 5
  TSH > ULN WITH FT3/FT4 TEST MISSING | 1 | 3
  TSH < LLN | 4 | 1
  TSH <LLN WITH TSH >= LLN AT BASELINE | 4 | 1
  TSH <LLN WITH ATLEAST ONE FT3/FT4 TEST VALUE > ULN | 3 | 1
  TSH <LLN WITH ALL OTHER FT3/FT4 TEST VALUES <= ULN | 1 | 0
  TSH < LLN WITH FT3/FT4 TEST MISSING | 0 | 0

16. Secondary Outcome: The Number of Participants With Abnormal Laboratory Values for Liver Tests
Description: The Number of Participants with Abnormal Laboratory Values for Liver Tests.
Time Frame: From first dose to 30 days post last dose (an average of 4 months up until a maximum of 7 months)
Population: All treated participants with at least one on treatment measurement.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Relapsed/Refractory Classic Hodgkin Lymphoma - Low Risk Relapse | Cohort 2: Relapsed/Refractory Classic Hodgkin Lymphoma - Standard Risk Relapse
Number analyzed (Participants) | 28 | 44
Participants
  ALT OR AST > 3XULN | 8 | 5
  ALT OR AST> 5XULN | 3 | 1
  ALT OR AST> 10XULN | 0 | 0
  ALT OR AST > 20XULN | 0 | 0
  TOTAL BILIRUBIN > 2XULN | 1 | 0
  ALT/AST ELEV>3XULN;TOTAL BILIRUBIN>2XULN IN 1 DAY | 0 | 0
  ALT/AST ELEV>3XULN;TOTAL BILIRUBIN>2XULN IN 30 DAYS | 0 | 0

17. Secondary Outcome: Number of Participants With Abnormal Vital Signs Reported as Adverse Events
Description: Temperature, blood pressure, and heart rate abnormalities reported as adverse events.
Time Frame: From first dose to 100 days after last dose of study therapy (assessed for an average of 7 months up until a maximum of 10 months).
Population: All treated participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Relapsed/Refractory Classic Hodgkin Lymphoma - Low Risk Relapse | Cohort 2: Relapsed/Refractory Classic Hodgkin Lymphoma - Standard Risk Relapse
Number analyzed (Participants) | 28 | 44
Participants
  Pyrexia | 7 | 23
  Tachycardia | 2 | 1
  Sinus Bradycardia | 0 | 2
  Hypertension | 0 | 4
  Hypotension | 0 | 6
  Orthostatic hypotension | 0 | 1

ADVERSE EVENTS:
Time Frame: Participants were assessed for All-Cause Mortality from first dose until study completion (assessed up to approximately 86 months). SAEs and Other AEs were assessed from first dose to 100 days after last dose of study therapy (assessed for an average of 7 months up until a maximum of 10 months).
Description: All-Cause Mortality, Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication. Data prespecified to be reported per treatment modality received in:
  1. induction phase and consolidation phase only for those who did not progress to intensification phase in each cohort.
  2. induction phase, intensification phase, and consolidation phase for those who proceeded to the intensification phase in each cohort.
Groups:
- Cohort 1: Relapsed/Refractory Classic Hodgkin Lymphoma - Low Risk Relapse (Nivo + Bv): Participants started in the induction phase and received nivolumab + brentuximab vedotin (N+Bv) for 2 cycles (6 weeks). Participants with radiographic progression, as assessed by Investigator at Cycle 2 entered follow-up. The rest of the participants continued in the induction phase and received 2 additional cycles of N+Bv study therapy (total 4 cycles = 12 weeks).
  - Participants who had a complete metabolic response (CMR) by BICR after a total of 4 cycles (12 weeks) of N+Bv received an additional 2 cycles of treatment of N+Bv (for a total of 6 cycles [18 weeks]), followed by Radiation Therapy (RT) (consolidation phase).
- Cohort 1: Relapsed/Refractory Classic Hodgkin Lymphoma - Low Risk Relapse (Nivo + Bv) + (Bv + B): Participants started in the induction phase and received nivolumab + brentuximab vedotin (N+Bv) for 2 cycles (6 weeks). Participants with radiographic progression, as assessed by Investigator at Cycle 2 entered follow-up. The rest of the participants continued in the induction phase and received 2 additional cycles of N+Bv study therapy (total 4 cycles = 12 weeks).
  * Participants who had a complete metabolic response (CMR) by BICR after a total of 4 cycles (12 weeks) of N+Bv received an additional 2 cycles of treatment of N+Bv (for a total of 6 cycles [18 weeks]), followed by Radiation Therapy (RT) (consolidation phase).
  * Participants without a CMR after 4 cycles of N+Bv, by BICR, entered the intensification phase and received 2 cycles of brentuximab + bendamustine (Bv+B); participants who achieved CMR after these 2 cycles proceeded with RT (consolidation phase).
  * Participants who had radiographic progression after Cycle 4 N+Bv, as assessed by BICR, or those who did not achieve CMR, by BICR, after 2 cycles of Bv+B were taken off study treatment and entered follow-up.
- Cohort 2: Relapsed/Refractory Classic Hodgkin Lymphoma - Standard Risk Relapse (Nivo + Bv): Participants started in the induction phase and received nivolumab + brentuximab vedotin (N+Bv) for 2 cycles (6 weeks). Participants with radiographic progression, as assessed by Investigator at Cycle 2 entered follow-up. The rest of the participants received 2 additional cycles of N+Bv study therapy (total 4 cycles = 12 weeks).
  - Participants who had complete metabolic response (CMR), by BICR, after a total of 4 cycles (12 weeks) of N+Bv proceeded with high-dose chemotherapy followed by an autologous stem cell transplant (HDCT/ASCT) (consolidation phase). Participants with CMR had the option to receive up to 2 additional cycles of N+Bv if their HDCT/ASCT was postponed for any reason.
- Cohort 2: Relapsed/Refractory Classic Hodgkin Lymphoma - Standard Risk Relapse (Nivo + Bv)+(Bv + B): Participants started in the induction phase and received nivolumab + brentuximab vedotin (N+Bv) for 2 cycles (6 weeks). Participants with radiographic progression, as assessed by Investigator at Cycle 2 entered follow-up. The rest of the participants received 2 additional cycles of N+Bv study therapy (total 4 cycles = 12 weeks).
  * Participants who had complete metabolic response (CMR), by BICR, after a total of 4 cycles (12 weeks) of N+Bv proceeded with high-dose chemotherapy followed by an autologous stem cell transplant (HDCT/ASCT) (consolidation phase). Participants with CMR had the option to receive up to 2 additional cycles of N+Bv if their HDCT/ASCT was postponed for any reason.
  * Participants without a CMR, by BICR, after 4 cycles of N+Bv received 2 cycles of brentuximab + bendamustine (Bv+B) (intensification phase).
  * Participants in CMR, by BICR, after 2 cycles of Bv+B received HDCT/ASCT (consolidation phase).
  * Participants without CMR by BICR could receive 2 additional cycles of Bv+B. If these participants attained CMR, they proceeded with HDCT/ASCT (consolidation phase).
  * Participants with CMR had the option to receive up to 2 additional cycles of B+Bv if their HDCT/ASCT was postponed.
  * Participants who had radiographic progression after Cycle 4 N+Bv, during study treatment or those who did not achieve CMR after final cycle of Bv+B were taken off study treatment and entered follow-up.
Arm/Group | Cohort 1: Relapsed/Refractory Classic Hodgkin Lymphoma - Low Risk Relapse (Nivo + Bv) | Cohort 1: Relapsed/Refractory Classic Hodgkin Lymphoma - Low Risk Relapse (Nivo + Bv) + (Bv + B) | Cohort 2: Relapsed/Refractory Classic Hodgkin Lymphoma - Standard Risk Relapse (Nivo + Bv) | Cohort 2: Relapsed/Refractory Classic Hodgkin Lymphoma - Standard Risk Relapse (Nivo + Bv)+(Bv + B)
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/6 | 0/33 | 1/11
Serious Adverse Events (participants affected / at risk) | 6/22 | 3/6 | 11/33 | 4/11
Other Adverse Events (participants affected / at risk) | 18/22 | 6/6 | 33/33 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Relapsed/Refractory Classic Hodgkin Lymphoma - Low Risk Relapse (Nivo + Bv) (N=22) | Cohort 1: Relapsed/Refractory Classic Hodgkin Lymphoma - Low Risk Relapse (Nivo + Bv) + (Bv + B) (N=6) | Cohort 2: Relapsed/Refractory Classic Hodgkin Lymphoma - Standard Risk Relapse (Nivo + Bv) (N=33) | Cohort 2: Relapsed/Refractory Classic Hodgkin Lymphoma - Standard Risk Relapse (Nivo + Bv)+(Bv + B) (N=11)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 2 | 3 | 3 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 1 | 1
Otitis media (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 1 | 0
Blood phosphorus increased (Investigations) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary veno-occlusive disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Relapsed/Refractory Classic Hodgkin Lymphoma - Low Risk Relapse (Nivo + Bv) (N=22) | Cohort 1: Relapsed/Refractory Classic Hodgkin Lymphoma - Low Risk Relapse (Nivo + Bv) + (Bv + B) (N=6) | Cohort 2: Relapsed/Refractory Classic Hodgkin Lymphoma - Standard Risk Relapse (Nivo + Bv) (N=33) | Cohort 2: Relapsed/Refractory Classic Hodgkin Lymphoma - Standard Risk Relapse (Nivo + Bv)+(Bv + B) (N=11)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 6 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 5 | 4
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 2 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 4 | 2
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 2
Tachycardia (Cardiac disorders) | 2 | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 2 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 1
Eye pain (Eye disorders) | 0 | 0 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 9 | 4
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 7 | 1
Coating in mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 4 | 0 | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 5 | 1 | 13 | 4
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 9 | 3 | 19 | 11
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 7 | 1
Vomiting (Gastrointestinal disorders) | 2 | 3 | 7 | 6
Asthenia (General disorders) | 4 | 1 | 1 | 1
Face oedema (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 4 | 2 | 7 | 1
Gait disturbance (General disorders) | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 1 | 1 | 1
Mucosal inflammation (General disorders) | 1 | 0 | 10 | 5
Non-cardiac chest pain (General disorders) | 1 | 0 | 1 | 1
Oedema peripheral (General disorders) | 0 | 0 | 2 | 0
Pyrexia (General disorders) | 1 | 2 | 17 | 5
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 2 | 1
Hypersensitivity (Immune system disorders) | 1 | 2 | 6 | 3
Infusion related hypersensitivity reaction (Immune system disorders) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 1
Epstein-Barr virus infection reactivation (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1 | 1
Otitis media (Infections and infestations) | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 3 | 1
Rhinitis (Infections and infestations) | 1 | 2 | 3 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 2 | 2
Urinary tract infection (Infections and infestations) | 2 | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 4 | 1 | 4 | 5
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Radiation associated pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Radiation skin injury (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 0
Vascular access site pruritus (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 5 | 2 | 2 | 3
Amylase increased (Investigations) | 1 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 3 | 2 | 3 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 1
Blood bilirubin increased (Investigations) | 2 | 0 | 0 | 0
Body temperature increased (Investigations) | 0 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 1
Heart rate increased (Investigations) | 0 | 1 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 1
Lipase decreased (Investigations) | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 2 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 1 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 2 | 0
Platelet count decreased (Investigations) | 0 | 0 | 4 | 2
Weight decreased (Investigations) | 1 | 0 | 2 | 1
White blood cell count decreased (Investigations) | 1 | 0 | 2 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 8 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hypouricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 5 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 2 | 2 | 2
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 4 | 1
Headache (Nervous system disorders) | 10 | 2 | 6 | 4
Presyncope (Nervous system disorders) | 1 | 0 | 2 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 3 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 2 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 2 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 8 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 4 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 4 | 1
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 1 | 5 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 3 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 3 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 0 | 2 | 3
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 1 | 6 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 3 | 1
Hypotension (Vascular disorders) | 0 | 0 | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-26): https://cdn.clinicaltrials.gov/large-docs/69/NCT02927769/Prot_SAP_000.pdf